CLINICAL TRIAL: NCT02210078
Title: Most Closely HLA Matched Allogeneic CMV Specific Cytotoxic T-Lymphocytes (CTL) to Treat CMV Infection After Hemapoietic Stem Cell Transplantation (HSCT)
Brief Title: Donor Cytomegalovirus-Specific Cytotoxic T-Lymphocytes in Treating Patients With a Persistent Cytomegalovirus Infection
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0657; NCI-2014-01990 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-0657 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2025-08

CONDITIONS: Cytomegaloviral Infection; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Cytomegalovirus Infections; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (allogeneic CMV-specific cytotoxic T-lymphocytes) (Experimental): Patients receive allogeneic cytomegalovirus-specific cytotoxic T-lymphocytes IV. Patients with partial response, stable disease, or progressive disease may receive an additional dose of allogeneic cytomegalovirus-specific cytotoxic T-lymphocytes at a minimum of 2 weeks from the first infusion.
  Interventions: Biological: Allogeneic Cytomegalovirus-Specific Cytotoxic T lymphocytes

INTERVENTIONS:
Biological: Allogeneic Cytomegalovirus-Specific Cytotoxic T lymphocytes — Given IV

SUMMARY:
This phase II trial studies how well donor cytomegalovirus-specific cytotoxic T-lymphocytes work in treating patients with a cytomegalovirus infection that has come back or has not gotten better despite standard therapy. White blood cells from donors who have been exposed to cytomegalovirus may be effective in treating patients with a cytomegalovirus infection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the efficacy, feasibility and safety of administering most closely human leukocyte antigen (HLA)-matched cytomegalovirus (CMV) specific cytotoxic T-lymphocytes (HMC-CTLs) generated by "gamma-catch" to mediate antiviral activity in hematopoietic stem cell transplantation (HSCT) recipients with CMV infections.

SECONDARY OBJECTIVE:

I. To assess the persistency of the administered HMC-CTLs generated by "gamma-catch" and their contribution immune reconstitution.

OUTLINE:

Patients receive allogeneic cytomegalovirus-specific cytotoxic T-lymphocytes intravenously (IV). Patients with partial response, stable disease, or progressive disease may receive an additional dose of allogeneic cytomegalovirus-specific cytotoxic T-lymphocytes at a minimum of 2 weeks from the first infusion.

After completion of study treatment, patients are followed up periodically for 12 months.

ELIGIBILITY:
Inclusion criteria:

Patients with or without a malignancy; and/or any type of autologous or allogeneic HSCT; and/or patients who are immunocompromised with CMV infection will be included.

Persistent CMV infection despite optimum anti-viral therapy

1. Patients with CMV disease: defined as the demonstration of CMV by biopsy specimen from visceral sites (by culture or histology) or the detection of CMV by culture or direct fluorescent antibody stain in bronchoalveolar lavage fluid in the presence of new or changing pulmonary infiltrates OR
2. Failure of antiviral therapy: defined as the continued presence of DNAemia (defined as >/= 137 copies/ml by PCR) for at least 2 weeks of CMV antiviral therapy OR

   1. Optimum therapy is defined as at least 14 days of therapy with Ganciclovir, Foscarnet, Cidofovir, or Valganciclovir for patients with disease or CMV viremia.
   2. Relapse while on CMV antiviral therapy defined as recurrence of DNAemia while being on at least 2 weeks of antiviral therapy OR
3. Patients who cannot tolerate standard anti-viral therapy and cannot continue anti-viral treatment due to side effect profile will be eligible independent of anti-viral therapy duration.

Clinical status at enrollment to allow tapering of steroids equal to or less than 0.5 mg/kg/day of prednisone.

Patients with chronic GVHD if on prednisone equal to or less than 0.5 mg/kg and not receiving second-line GVHD treatments like Pentostatin, Infliximab, Etanercept, etc.

Written informed consent and/or signed assent line from patient, parent or guardian.

Written informed consent from patient or legally authorized representative (LAR). Patients with cognitive impairment are eligible.

* Negative pregnancy test in female patients of childbearing potential.
* Patients ≥ 2 years.
* English and non-English speaking patients are eligible.
* Patients enrolled on this study may be enrolled on other IND studies at the discretion of the PI.

Exclusion criteria:

* Patients receiving prednisone >0.5 mg/kg/day at time of enrollment, or have received ATG, donor lymphocyte infusion (DLI) or Campath within 28 days of enrollment.
* Patients with other uncontrolled infections. For bacterial infections, patients must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to enrollment. For fungal infections patients must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection for 1 week prior to enrollment. Progressing infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection. Patients with ongoing viral infections are excluded.
* Patients with active acute GVHD grades II-IV.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-02-19 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Success, defined as R1 and R2 without treatment failure | Up to 4 weeks after second CTL infusion
  The best outcome is defined as R1 = in complete response (CR) for 4 consecutive weeks, starting at week 2, without the need for a second cytotoxic T-lymphocyte (CTL) infusion. The second best outcome is defined as R2 = not in CR at week 2, 3, or 4, but in CR or partial response (PR) 4 weeks after the second CTL infusion.

SECONDARY OUTCOMES:
Overall survival time | Up to 12 months
  Will be analyzed as a function of patient covariates using standard statistical methods, including Bayesian survival regression analysis and ordinal regression. Unadjusted event time distributions will be estimated using the Kaplan-Meier method.
Disease-free survival time | Up to 12 months
  Will be analyzed as a function of patient covariates using standard statistical methods, including Bayesian survival regression analysis and ordinal regression. Unadjusted event time distributions will be estimated using the Kaplan-Meier method.
Graft-versus-host disease | Up to 12 months
  Will be analyzed as a function of patient covariates using standard statistical methods, including Bayesian survival regression analysis and ordinal regression.
Secondary graft failure | Up to 12 months
  Will be analyzed as a function of patient covariates using standard statistical methods, including Bayesian survival regression analysis and ordinal regression.

CONTACTS AND LOCATIONS:
Overall Officials: Betul Oran, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org